CLINICAL TRIAL: NCT07177378
Title: Management of Medication Related Osteonecrosis of the Jaws Using Piezosurgery With Simultaneous Double Periosteal Flap Closure
Brief Title: Management of Medication Related Osteonecrosis of the Jaws With Double Periosteal Flap Closure
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, mona samy sheta, lecturer of oral and maxillofacial surgery, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1981
Record Dates: First submitted 2025-09-15; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Osteomyelitis of Jaw
Keywords: medication related osteonecrosis; mandible; piezosurgery

STUDY DESIGN:
Intervention Model Description: patient with medication related osteonecrosis of the mandible underwent surgical debridement and closure using double periosteal flap
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- management of medication related osteonecrosis of the jaw (Experimental): The buccal mucoperiosteal flap was elevated to expose the area of osteonecrosis in the mandible. it was debrided using piezosurgery then closure was achieved using double periosteal flap
  Interventions: Device: management of medication related osteonecrosis of the jaw

INTERVENTIONS:
Device: management of medication related osteonecrosis of the jaw — after buccal flap reflection, the bone osteonecrosis was debrided using piezosurgery. the buccal mucoperiosteal flap was dissected to two layers first, the periosteal layer was based superiorly and the mucosal flap to achieve double layers closure.

SUMMARY:
20 patients with MRONJ underwent surgical debridement using piezosurgery then closure using double periosteal flap

DETAILED DESCRIPTION:
20 patients with MRONJ underwent surgical debridement, crestal incision and oblique releasing incision were performed to expose the area of osteomyelitis, then squesterum was removed using piezosurgery. After complete debridement, the periosteal layer was dissected from mucoperiosteal buccal flap and based superiorly, then turn upward to be sutured to the lingual flap followed by suturing of buccal flap to achieve double layers closure

ELIGIBILITY:
Inclusion Criteria:

* patients with MRONJ

Exclusion Criteria:

* patients had a history of radiotherapy Patients need only conservative treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
evaluation of pain | one month
  visual analog scale (VAS), with 0 indicating no pain and 10 indicating the most severe pain.
wound healing | one -3 months
  the wound healing index (WHI) which scored soft tissue healing according to the following criteria: score 1 = uneventful healing with no gingival edema, erythema, suppuration, patient discomfort, or flap dehiscence; score 2 = uneventful healing with slight gingival edema, erythema, patient discomfort, or flap dehiscence, but no suppuration; and score 3 = poor wound healing with significant gingival edema, erythema, patient discomfort, flap dehiscence, or any suppuration

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt